CLINICAL TRIAL: NCT05749978
Title: Effects of Postural Adjustment on Hemodynamics in Patients Undergoing Prone Spine Surgery Under General Anesthesia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhuan Zhang (Other)
Responsible Party: Sponsor-Investigator, Zhuan Zhang, Principal Investigator, Yangzhou University
Organization: Yangzhou University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 20230218
Record Dates: First submitted 2023-02-18; First posted 2023-03-01 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-01

CONDITIONS: Asana Adjustment
Keywords: Trendelenburg position; Prone Position; Hemodynamics; Intra-abdominal pressure; Cardiac output

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trendelenburg position (Experimental)
  Interventions: Behavioral: Asana adjustment
- Procumbent (No Intervention)

INTERVENTIONS:
Behavioral: Asana adjustment — Adjust the operating table to 15° head height and foot low in advance. The patient is then slowly turned over from the transport table to the operating table and completed in the prone position. After the patient's hemodynamic stability is smooth, adjust the operating table to the level.
  Arms: Trendelenburg position

SUMMARY:
The prone position is a special position often used for spinal surgery. As a special position of general anesthesia, after induction of general anesthesia, severe hemodynamic fluctuations often occur when the supine position is changed to the prone position, which seriously affects the patient's circulatory and respiratory functions.

ELIGIBILITY:
Inclusion Criteria:

1. Prone spine surgery after general anesthesia is planned.
2. Age 18~85 years old.
3. ASA grade I or II.
4. BMI18.3-30kg/m2

Exclusion Criteria:

1. Unstable angina or myocardial infarction, coronary heart disease, congestive heart failure, structural heart disease, arrhythmia within 6 months;
2. Increased intracranial pressure and central nervous system injury or disease;
3. Severe hypertension
4. Patients with other diseases affecting their own circulatory system.
5. Have or have a history of severe mental disorders;
6. Bleeding volume >600ml or intraoperative blood transfusion treatment.
7. Severe liver and kidney insufficiency

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-10-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in Blood pressure | Preoperatively,5 minute after anesthesia induction,Immediately before the prone position, Immediately after the prone position,1 minute after prone position, 3 minute after prone position,10 minute after prone position,Half an hour after prone position
  Hemodynamics
Changes in the level of Cardiac output | Preoperatively,5 minute after anesthesia induction,Immediately before the prone position, Immediately after the prone position,1 minute after prone position, 3 minute after prone position,10 minute after prone position,Half an hour after prone position
  Cardiac output

SECONDARY OUTCOMES:
Intra-abdominal pressure level | Preoperatively,5 minute after anesthesia induction,Immediately before the prone position, Immediately after the prone position,1 minute after prone position, 3 minute after prone position,10 minute after prone position,Half an hour after prone position
  Intra-abdominal pressure
Vasoactive drugs | Intraoperatively
  Vasoactive drug dosage

CONTACTS AND LOCATIONS:
Locations (1):
- the Affiliated Hospital of Yangzhou University, Yangzhou University, Yangzhou, Jiangsu, China